CLINICAL TRIAL: NCT01768299
Title: Medical Abortion With Mifepristone + Misoprostol (13 - 22 Weeks): A Double-blind Randomized-controlled Trial
Brief Title: Medical Abortion With Mifepristone + Misoprostol (13 - 22 Weeks)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1008
Record Dates: First submitted 2013-01-11; First posted 2013-01-15 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Complete Uterine Evacuation After Use of Study Drugs
Keywords: abortion; medical abortion; mifepristone; misoprostol
MeSH Terms: interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mifepristone at home 24 hours before miso dosing starts (Experimental): All women will receive study packet one containing mifepristone to swallow at home on study day 1. They will be told to return to the hospital for induction and will be scheduled to return to the hospital 24 hours later. Upon their return, they will be hospitalized and receive another study packet containing a placebo. Simultaneously, they will receive one dose of 400 mcg buccal misoprostol. Women will remain hospitalized and receive repeated doses of 400 mcg buccal misoprostol every three hours.
  Participants will receive up to eight doses of misoprostol (e.g. 3200 mcg misoprostol) over 24 hours. Misoprostol dosing will stop when both the fetus and placenta are expelled.
  Interventions: Drug: Mifepristone
- Mifepristone and first dose of misoprostol simultaneously. (Experimental): Will receive study packet one containing placebo to swallow at home on study day 1. They will be told to return to the hospital for induction and will be scheduled to return to the hospital 24 hours later. Upon their return, they will be hospitalized and receive another study packet containing mifepristone. Simultaneously they will receive one dose of 400 mcg buccal misoprostol. Women will remain hospitalized and receive repeated doses of 400 mcg buccal misoprostol every three hours.
  Participants will receive up to eight doses of misoprostol (e.g. 3200 mcg misoprostol) over 24 hours. Misoprostol dosing will stop when both the fetus and placenta are expelled. The procedure will be considered complete once both the fetus and placenta are expelled.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Mifepristone — 200 mg oral Mifepristone 24 hours before 400 mcg buccal misoprostol
  Arms: Mifepristone at home 24 hours before miso dosing starts
Drug: Misoprostol — 200 mg oral Mifepristone simultaneously 400 mcg buccal misoprostol
  Arms: Mifepristone and first dose of misoprostol simultaneously.

SUMMARY:
A double-blind randomized controlled trial to compare a shorter interval between the administration of mifepristone and misoprostol (simultaneous administration compared to 24hours from administration of mifepristone to receipt of the first dose of misoprostol) for termination of pregnancy up to 13-22 weeks of gestation. The investigators hypothesize that a shortened interval may achieve comparable efficacy in terminating pregnancy, whilst reducing the duration of the procedure and in turn, the duration of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Closed cervical os and no vaginal bleeding
* Live fetus at time of presentation for service
* No contraindications to medical abortion and study procedures, according to provider
* Able to consent to participate in the study, either by reading consent document or by having consent document read to her and sign informed consent
* Willing to follow study procedures

Exclusion Criteria:

* Known previous transmural uterine incision
* > 5 parity
* Signs and symptoms of infection
* Any contraindications to vaginal delivery, including placenta previa
* Presentation in active labor (defined as moderate to severe contractions every 10 minutes or less)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2013-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Proportion of women who have had a complete uterine evacuation within 24 hours using study drug without recourse to any additional intervention. | Within 1 week
  Defined as complete evacuation of fetus and placenta using study drug without recourse to any additional intervention.

SECONDARY OUTCOMES:
Induction to abortion interval | Within 1 week
  Defined as time elapsed between administration of the first misoprostol dose until expulsion of the fetus and placenta.
Women's acceptability of the assigned method. | Within 1 week
Rate of fetal expulsion | Within 1 week
  Defined as fetal expulsion with study drug alone.
Provision of additional interventions | Within 1 week
  For example: Uterine massage, Manual removal, Sponge forceps, D&C or D&E, Repeat medical abortion drugs
Time interval from the mifepristone dose to abortion | Within 1 week
  Defined as length of time from initiation of mifepristone to complete abortion achieved.
Total dose of misoprostol administered | Within 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Blum, MPH, Principal Investigator — Gynuity Health Projects; Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects; Dina Abbas, MPH, Principal Investigator — Gynuity Health Projects; Nguyen thi Ngoc, MD, Principal Investigator — Hung Vuong Hospital
Locations (3):
- Vietnam (3):
  - Binh duong Obstetrics and Newborn Hospital, Ho Chi Minh City, Binh Duong Province
  - National Ob-Gyn Hospital, Hanoi
  - Hung Vuong Hospital, Ho Chi Minh City

REFERENCES:
- [Derived] Abbas DF, Blum J, Ngoc NT, Nga NT, Chi HT, Martin R, Winikoff B. Simultaneous Administration Compared With a 24-Hour Mifepristone-Misoprostol Interval in Second-Trimester Abortion: A Randomized Controlled Trial. Obstet Gynecol. 2016 Nov;128(5):1077-1083. doi: 10.1097/AOG.0000000000001688. PMID 27741182